CLINICAL TRIAL: NCT00922233
Title: Pericoital Oral Contraception With Levonorgestrel: A Prospective, Open-Label, Single Arm, Multicenter Study to Evaluate Efficacy, Safety and Acceptability
Brief Title: Pericoital Oral Contraception With Levonorgestrel
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: FHI 360 (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 10139
Record Dates: First submitted 2009-06-10; First posted 2009-06-17 (Estimated); Results first posted 2013-10-29 (Estimated); Last update posted 2013-10-29 (Estimated); Status verified 2013-08

CONDITIONS: Healthy
Keywords: Contraception
MeSH Terms: interventions — Levonorgestrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Levonorgestrel (Experimental): 0.75 mg of levonorgestrel within 24 hours of sex
  Interventions: Drug: levonorgestrel

INTERVENTIONS:
Drug: levonorgestrel — oral contraceptive pills

SUMMARY:
A prospective, open-label, single arm, multicenter study to evaluate efficacy, safety and acceptability of pericoital oral contraception with levonorgestrel

DETAILED DESCRIPTION:
This is a prospective, open-label, single arm, multicenter study to evaluate efficacy, safety and acceptability of pericoital oral contraception with levonorgestrel (LNG). The objectives of the study as stated in the study protocol are as follows:

* To evaluate the efficacy of the study regimen among women who have sex 1-4 days a month and who are relying on the study regimen as their primary method of contraception
* To evaluate the safety of this regimen, with particular emphasis on its effects on vaginal bleeding patterns and anemia
* To evaluate the acceptability of the regimen The study will enroll fertile women of reproductive age who have sex up to 6 days a month, are at low risk for sexually transmitted infections (STIs), have no contraindications to progestin-only oral contraceptives,have no serious contraindications to pregnancy, and are willing to use an investigational method of contraception as their only contraceptive method for 6.5 months (each tablet contains 0.75 mg LNG to be used after every sex act).

ELIGIBILITY:
Inclusion Criteria:

Each woman enrolled in the trial must meet the following inclusion criteria:

* Competent to provide informed consent to participate in the trial and has done so.
* At least the minimum age is 18 to 45 years old.
* Had sex 1 to 4 days in past month and expects to continue at that frequency for the next 6.5 months.
* At low risk for sexually transmitted infection (STI), operationally meaning that neither she nor her partner to her knowledge has had any of the following:

  * More than one sexual partner currently or any expectation of having more than one sexual partner in the next 6.5 months
  * Diagnosis of human immunodeficiency virus (HIV) infection, hepatitis B or hepatitis C
  * Treatment for a STI within the past 6 months, excluding recurrent genital herpes or condyloma
  * Sharing of illicit injection drug equipment ever in the past.
* Willing to use the study regimen as her only contraceptive method for the next 6.5 months (except that she may also use condoms if needed for protection from STIs).
* Wants to avoid pregnancy for at least the next 6.5 months.
* Willing to accept an uncertain risk of pregnancy during the study.
* Gives correct answers to the informed consent quiz.
* Willing and able to follow all study requirements.

Exclusion Criteria:

To be eligible for enrollment, a woman must not meet any of the following exclusion criteria:

* Pregnant as verified by a pregnancy test at enrollment.
* Has an indication of current subfecundity, specifically:

  * Her last pregnancy ended within the last 8 weeks, or she has had fewer than two menstrual periods since resolution of last pregnancy
  * She has not had normal monthly menses for the past 2 months
  * She is currently breastfeeding
  * She has used any hormonal contraceptive other than emergency contraceptive pills since the onset of her last menstrual period
  * Has received an injection of a long term injectable contraceptive in the last 9 months
  * Currently has an intrauterine device
  * Has had a sterilization procedure or ectopic pregnancy
  * Has been diagnosed by a clinician as having a fertility problem
  * Her partner has had a sterilization procedure or infertility diagnosis, to her knowledge.
* She currently has known contraindications to progestin-only pills, specifically including the following conditions:

  * Unexplained abnormal vaginal bleeding
  * Deep venous thrombosis or pulmonary embolus
  * Active viral hepatitis
  * Decompensated cirrhosis
  * Liver tumor
  * History of breast cancer within the past 5 years.
* Has a breast mass on examination.
* Has a personal or family history suggestive of predisposition to thrombosis.
* Has a serious contraindication to pregnancy (medical condition or use of chronic medication such as isotretinoin or thalidomide).
* Taking drugs that are known to interact with progestins (such as rifampicin or anticonvulsant medications).
* Has previously participated in this study.
* Currently participating in another medical research study.
* The site investigator or designee perceives another reason to exclude her from the trial.

Max Age: 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 72 (Actual)
Dates: Start 2010-01; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vera Halpern, MD, Principal Investigator — FHI 360
Locations (4):
- United States (3):
  - Planned Parenthood of the Rocky Mountains, Denver, Colorado
  - Planned Parenthood Gulf Coast, Inc., Houston, Texas
  - Planned Parenthood Association of Utah, Salt Lake City, Utah
- CEMICAMP, Campinas, Campinas, Brazil

REFERENCES:
- [Derived] Taylor DJ, Lendvay A, Halpern V, Bahamondes LG, Fine PM, Ginde SY, Wheeless A, Raymond EG. A single-arm study to evaluate the efficacy, safety and acceptability of pericoital oral contraception with levonorgestrel. Contraception. 2014 Mar;89(3):215-21. doi: 10.1016/j.contraception.2013.11.013. Epub 2013 Nov 26. PMID 24388695

RESULTS

PARTICIPANT FLOW:
Groups:
- Levonorgestrel: Only one study arm. All women were assigned to take 0.75 mg oral contraceptive pills (levonorgestrel) within 24 hours of engaging in sex.
Period: Overall Study
Arm/Group | Levonorgestrel
Started | 72
Completed | 68
Not Completed | 4

BASELINE CHARACTERISTICS:
Groups:
- Levonorgestrel: 0.75 mg levonorgestrel oral contraceptive pills (levonorgestrel) : oral contraceptive pills
Arm/Group | Levonorgestrel
Number analyzed (Participants) | 72
Age Continuous [Mean (Standard Deviation); unit: years] | 32.4 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72
  Male | 0
Region of Enrollment [Number; unit: participants]
  Africa | 72

OUTCOME MEASURES:

1. Primary Outcome: Efficacy: the Pearl Index (Number of Pregnancies Per 100 Woman-years) in the Primary Evaluable Population (18-35)
Description: Participants were followed for 6.5 months.Pearl Index in the 18-35 year population was collected excluding months in which barrier methods, condoms, or emergency contraception were used unless the subject conceived
Time Frame: 6.5 months
Measure: Number; unit: pregnancies per 100 woman years
Groups:
- Levonorgestrel: 0.75 mg levonorgestrel oral contraceptive pills
Arm/Group | Levonorgestrel
Number analyzed (Participants) | 68
pregnancies per 100 woman years | 22.4

2. Secondary Outcome: Acceptability Based on Bleeding Patterns Reported
Description: Number of participants who reported bleeding patterns were acceptable and would therefore use Levonorgestrel
Time Frame: 6.5 months
Population: A total of 56 women reported on their bleeding patterns, of these, 43 found it acceptable. Numbers reported in the participant Flow module, represent the total enrolled and the maximum number available for evaluation. Not all the enrolled participants could be analyzed for every outcome measure.
Measure: Number; unit: participants
Groups:
- Levonorgestrel Arm: Only one study arm. All women were assigned to take 0.75 mg oral contraceptive pills (levonorgestrel) within 24 hours of engaging in sex.
Arm/Group | Levonorgestrel Arm
Number analyzed (Participants) | 56
participants | 43

3. Primary Outcome: Participant Report of Adverse Events.
Description: Safety data includes data from each subject up to two weeks after her last use of the study tablets as well as all events deemed related to study product, regardless of date last tablet was taken
Time Frame: 6.5 months
Population: A total of 58 women documented use of product on coital diaries and are included in the User Population for primary safety analysis. Numbers reported in the participant Flow module, represent the total enrolled and the maximum number available for evaluation. Not all the enrolled participants could be analyzed for every outcome measure.
Measure: Number; unit: adverse events
Arm/Group | Levonorgestrel Arm
Number analyzed (Participants) | 58
adverse events | 45

ADVERSE EVENTS:
Arm/Group | Levonorgestrel Arm
Serious Adverse Events (participants affected / at risk) | 0/72
Other Adverse Events (participants affected / at risk) | 28/72
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Levonorgestrel Arm (N=72)
anemia (Blood and lymphatic system disorders) | 10 (11)
nausea (Gastrointestinal disorders) | 2 (2)
vomiting (Gastrointestinal disorders) | 1 (1)
irritability (General disorders) | 1 (1)
hypersensitivity (Immune system disorders) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
chlamydial infection (Infections and infestations) | 1 (1)
ear infection (Infections and infestations) | 1 (1)
influenza (Infections and infestations) | 1 (1)
rhinitis (Infections and infestations) | 1 (1)
sinusitis (Infections and infestations) | 1 (1)
tonsilitis (Infections and infestations) | 1 (1)
upper respiratory tract infection (Infections and infestations) | 2 (2)
urinary tract infections (Infections and infestations) | 1 (1)
vaginal candidiasis (Infections and infestations) | 5 (5)
pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
headache (Nervous system disorders) | 3 (4)
dysuria (Renal and urinary disorders) | 1 (1)
cervical dysplasia (Reproductive system and breast disorders) | 1 (1)
decereased libido (Reproductive system and breast disorders) | 1 (1)
vaginal discharge (Reproductive system and breast disorders) | 3 (3)
cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
dermititis allergic (Skin and subcutaneous tissue disorders) | 1 (1)
seborrhea (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No